CLINICAL TRIAL: NCT01553838
Title: A Prospective Study to Evaluate MRI Guided Biopsy Compared With Transrectal Ultrasound Guided Biopsy of the Prostate in Men With Increased PSA Values
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Sponsor
Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 002
Record Dates: First submitted 2012-03-01; First posted 2012-03-14 (Estimated); Last update posted 2014-08-19 (Estimated); Status verified 2012-03

CONDITIONS: Prostate Cancer
Keywords: prostate biopsy; MRI guided biopsy; TRUS guided biopsy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sequentially MRI guided and TRUS guided biopsy (Experimental): Targeted MRI guided biopsy according to findings in a multiparametric MRI followed by transrectal guided biopsy
  Interventions: Device: MRI guided prostate biopsy and TRUS guided biopsy

INTERVENTIONS:
Device: MRI guided prostate biopsy and TRUS guided biopsy — MRI guided prostate biopsy

SUMMARY:
The purpose of this study is to determine whether MRI guided prostate biopsy achieves higher prostate cancer detection rates compared with transrectal ultrasound guided prostate biopsy in patients with increased PSA values > 4.0 ng/ml.

ELIGIBILITY:
Inclusion Criteria:

* PSA > 4.0 ng/ml
* written informed consent
* age >18

Exclusion Criteria:

* patients with prostate cancer
* patients with prior prostate biopsy
* patients with contraindications against MRI or biopsy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2012-01; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Prostate cancer detection rate | 3 years

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a measure of Safety and Tolerability | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Christian Arsov, MD, Principal Investigator — Department of Urology, University of Duesseldorf
Locations (1):
- Department of Urology, Düsseldorf, Germany